CLINICAL TRIAL: NCT04796454
Title: Pamiparib and Low Dose Temozolomide In Patients With Platinum Sensitive Biliary Tract Cancer
Acronym: PAMICC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1912-GITCG
Record Dates: First submitted 2021-02-01; First posted 2021-03-12 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Platinum-Sensitive Biliary Tract Cancer
Keywords: Pamiparib; Biliary Tract Cancer; Temozolomide
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cisplatin; Gemcitabine; Oxaliplatin; pamiparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CisGem/GemOx (Active Comparator): Cisplatin/Gemcitabine (3-week cycle):
  * Cisplatin IV 25 mg/m² d1 and day8
  * Gemcitabine 1000 mg/m² d1 and d8
  This treatment regimen will be given until documented disease progression, unacceptable toxicity, or patient refusal, for a maximum of 2 years.
  In case of unacceptable toxicity the CisGem regimen can also be switched to a GemOx regimen (4-week cycle):
  * Oxaliplatin IV 100 mg/m² d1 and day15
  * Gemcitabine 1000 mg/m² d1 and d15
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Oxaliplatin
- PamTMZ (Experimental): Pamiparib + temozolomide (4-week cycle):
  Pamiparib 60 mg PO twice a day d1-d28 Temozolomide 60 mg PO daily d1-d7
  This treatment regimen will be given until documented disease progression, unacceptable toxicity, or patient refusal, for a maximum of 2 years.
  Interventions: Drug: Pamiparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Cisplatin — Cisplatin IV 25 mg/m² on d1 and d8 - always combined with Gemcitabine; maximum treatment 2 years
  Arms: CisGem/GemOx
Drug: Gemcitabine — Gemcitabine IV 1000 mg/m² on d1 and d8 if in combination with Cisplatin; Gemcitabine IV 1000 mg/m² on d1 and d15 if in combination with Oxaliplatin; maximum treatment 2 years
  Arms: CisGem/GemOx
Drug: Oxaliplatin — Oxaliplatin IV 100 mg/m² on d1 and d15 - always combined with Gemcitabine; maximum treatment 2 years
  Arms: CisGem/GemOx
Drug: Pamiparib — Pamiparib 60 mg PO twice a day from d1 to day28 in a 4-week cycle - always combined with Temozolomide; until progression or maximum treatment 2 years
  Arms: PamTMZ
Drug: Temozolomide — Temozolomide 60 mg PO once a day from d1 to d7 in a 4-week cycle - always combined with Pamiparib; until progression or maximum treatment 2 years
  Arms: PamTMZ

SUMMARY:
The main objective of this trial is to evaluate the activity of pamiparib plus low dose TMZ as maintenance treatment in improving progression free survival (PFS) in patients with advanced BTC who have received first line platinum-based chemotherapy.

The primary objective is to test with a one-sided type I error of 10% whether pamiparib plus low dose TMZ as maintenance treatment increases PFS according to RECIST (version 1.1) in the entire study population as compared to standard treatment with Cisplatin-Gemcitabine chemotherapy regimen (or Gemcitabine-Oxaliplatin if cisplatin is contra-indicated).

This is an open label randomized controlled multi-center phase II trial.

Patients must meet all the criteria to be eligible. Eligible patients will be centrally randomized between the two arms in a 1:1 ratio. Randomization will be stratified by the following factors:

* Tumour response CR/PR vs SD vs non-measurable/non-PD after previous platinum-based chemotherapy as confirmed by central review
* Tumour location (intrahepatic bile ducts vs. gallbladder vs. perihilar bile ducts and distal bile duct and /ampulla of Vater tumours).

Patients will receive treatment until progression or for a maximum period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance status 0-1
* Histologically-proven diagnosis of biliary tract adenocarcinoma(BTC): intrahepatic-, perihilar or distal bile duct adenocarcinoma, gallbladder adenocarcinoma or ampulla of Vater adenocarcinoma, as per AJCC 8th Edition.

Note: patients with 'cholangiocarcinoma not otherwise specified but not intrahepatic' can be enrolled;

* Locally advanced, recurrent or metastatic disease stage
* Prior treatment: One maximum prior line of systemic treatment: Platinum-based treatment (CisGem or GemOx in case of contraindication to cisplatin) duration up to 18 weeks (4-6 cycles) for locally advanced or metastatic disease

  * Patients should have completed at least 80 % of the planned dose
  * Patients should have received the last dose at the maximum 2 weeks before study registration
* Non-progressive, measurable or non-measurable disease after platinum-based treatment as assessed by CT scan/MRI (RECIST 1.1), for central review
* Non-measurable disease is allowed if non PD as per RECIST 1.1 as confirmed by central review, and no radiological nor clinical progression as assessed by the investigator. In the absence of measurable disease, progression is defined as a change in non-measurable disease comparable in magnitude to the increase that would be required to declare PD for measurable disease or appearance of new metastatic lesions (RECIST 1.1).
* Normal 12-lead ECG (patients with abnormal ECG will be eligible if changes are not considered clinically significant by the local investigator)
* Adequate organs and hematologic function:
* Hemoglobin ≥ 9 g/dL (prior transfusions are allowed if they have been done ≥ 3-4 days before testing the haemoglobin Hb)
* White blood cell (WBC) ≥ 3.0 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN), except in subjects with suspected or established diagnosis with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN.
* ALT (or AST) & alkaline phosphatase ≤ 3 x ULN; ≤ 5 x ULN in case of liver metastases
* Serum albumin ≥ 2.5 g/dL
* Estimated glomerular filtration rate (eGFR) according to MDRD should be >50ml/min
* International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants
* The following local treatment modalities are allowed prior to enrollment within the rules described (provided there has been a full recovery):

  * Surgery: patients may have undergone a non-curative operation (i.e., R2 resection [with macroscopic residual disease] or palliative bypass surgery only), performed at least 28 days before enrolment/randomization
  * Radiotherapy: patients may have received prior radiotherapy (with or without radiosensitising low-dose chemotherapy) for localised disease, provided the patient has fully recovered and at least 28 days have elapsed since the RT…and the measurable disease is outside of the previously-treated area
  * Photodynamic therapy (PDT) for localized disease only with no evidence of metastatic disease - patients may have received prior PDT, provided the patient has fully recovered and at least 28 days have elapsed since the PDT and the measurable disease is outside of the previously-treated area
  * Other previous localised treatments targeting intrahepatic lesions such as selective internal radiation therapy (SIRT), transarterial chemoembolisation (TACE) and radiofrequency ablation (RFA) are allowed, provided the patient has finished it at least 28 days prior to enrolment/randomization, with full recovery and the measurable disease is outside of the previously-treated area
* Any toxicity from CisGem/GemOx should be resolved, except for alopecia (any grade), grade 1 fatigue, grade 1 anorexia, grade 1 peripheral neurotoxicity, and grade 1 ototoxicity
* If clinically indicated, adequate biliary drainage or stent insertion should have been performed and patient should have fully recovered according to the treating physician
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression or other reasons.

* Women and men of childbearing / reproductive potential should use highly effective birth control measures, during the study treatment period and for at least 6 months after the last dose of treatment, as per CTFG guidelines
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Non-sterile males must use contraception during treatment and for 6 months after the last dose
* Non-sterile males must avoid sperm donation for the duration of the study and for at least 6 months after the last dose of study treatment.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Patients with squamous, all mixed with non-adenocarcinoma types (eg with neuroendocrine, hepatocellular, squamous, adenosquamous and medullar carcinoma)
* Prior therapy for BTC with an IDH 1 or 2 inhibitor or any other monoclonal antibodies
* Subjects with pleural effusion, pericardial effusion, or ascites with symptoms uncontrolled by medication or who require current drainage procedures (once monthly or more frequently).
* Central nervous system metastases or leptomeningeal spread of disease.
* Patients who are currently participating and receiving study therapy or have participated in a study with an investigational agent and received study therapy or used an investigational device wit weeks prior to enrolment/randomization.
* Patients with a previously treated malignancy are eligible to participate if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease. Exceptions: patients with currently treated basal cell, squamous cell carcinoma of the skin, localized treated low Gleason score prostate carcinoma (ie, resected prostate cancer staged pT1-2 with Gleason Score ≤ 6 and postoperative PSA < 0.5 ng/ml), or in-situ carcinoma of the cervix are eligible.
* Inability to swallow and/ or retain oral tablets
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Serious infection requiring oral or IV antibiotics within 7 days prior to registration
* Known contraindication to either cisplatin, oxaliplatin, gemcitabine
* Known contraindication to imaging tracer or any product of contrast media and CT/MRI contraindications
* Hypersensitivity to the active substance temozolomide or to any of the excipients listed in the SmPC.
* Hypersensitivity to dacarbazine (DTIC).
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Has known history or current evidence of HIV
* Has known history of chronic Hepatitis B or C or current evidence of active Hepatitis B or Hepatitis C.

Note: patient will be eligible if

* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 36 months from randomization
  Progression-free survival according to RECIST v1.1 from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Incidence of adverse events (safety and toxicity) | 25 months from randomization
  Assessment of adverse events according to CTCAE v5.0 - From date of randomization until the date of end of treatment visit or date of death from any cause, whichever came first, assessed up to 25 months
PFS as per central review | 36 months from randomization
  PFS as per central review assessment from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
overall survival (OS) | 36 months from randomization
  Overall survival from date of randomization until the date of end of treatment visit or date of death from any cause, whichever came first, assessed up to 36 months
Best overall response | 36 months from randomization
  Best overall response according to RECIST v1.1 from date of randomization until the date of end of treatment visit or date of death from any cause, whichever came first, assessed up to 36 months
Global Health Status/Quality of Life/physical functioning | 6 months from randomization
  Global Health Status/Quality of Life/physical functioning assessed with EORTC QLQ-30 questionnaire from date of randomization until 6 months thereafter or until date of death from any cause, whichever came first.
  This instrument is composed of multi-item and single-item scales. These include five functional scales (physical, role, emotional, social, and cognitive), three symptom (fatigue, nausea and vomiting and pain) and a global health status/QoL scale and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties).
  The scales range from 0 to 100 with the worst score being 0 for functioning scales and 100 for symptom scales.
Jaundice scale | 6 months from randomization
  Jaundice scale assessed with EORTC QLQ-BIL21 questionnaire from date of randomization until 6 months thereafter or until date of death from any cause, whichever came first.
  The Cholangiocarcinoma and Gallbladder Cancer Module (QLQ-BIL21) is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-BIL21 incorporates five multi-item scales to assess eating, jaundice, tiredness, pain and anxiety. In addition, three single items assess treatment side-effects, drainage bags/tubes and weight loss.
  The scales range from 0 to 100.